CLINICAL TRIAL: NCT01732822
Title: A Randomized, Double-blind, Parallel Group, Multicentre Phase IIIb Study to Compare Ticagrelor With Clopidogrel Treatment on the Risk of Cardiovascular Death, Myocardial Infarction and Ischemic Stroke in Patients With Established Peripheral Artery Disease (EUCLID Examining Use of tiCagreLor In paD)
Brief Title: A Study Comparing Cardiovascular Effects of Ticagrelor and Clopidogrel in Patients With Peripheral Artery Disease
Acronym: EUCLID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5135C00001; 2011-004616-36 (EudraCT Number)
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-09

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral artery disease Atherothrombotic events Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Ticagrelor 90 mg bd (and Clopidogrel placebo od) taken orally as tablets
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Clopidogrel 75 mg od (and Ticagrelor placebo bd) taken orally as tablets
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90 mg bd (and Clopidogrel placebo od) taken orally as tablets
  Other Names: Brilinta/Brilique
  Arms: Ticagrelor
Drug: Clopidogrel — Clopidogrel 75 mg od (and Ticagrelor placebo bd) taken orally as tablets
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to compare the effects of ticagrelor and clopidogrel in patients with Peripheral Artery Disease.

DETAILED DESCRIPTION:
A randomized, double-blind, parallel group, multicentre phase IIIb study to compare ticagrelor with clopidogrel treatment on the risk of cardiovascular death, myocardial infarction and ischemic stroke in patients with established Peripheral Artery Disease (EUCLID Examining Use of tiCagreLor In paD)

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients 50 years old or older Symptomatic peripheral artery disease

Exclusion Criteria:

* Patients needing dual anti-platlet drug treatment before start of study Planned revascularisation or amputation
* Patients with known bleeding disorders
* Patients with a history of intracranial bleed
* Patients considered to be at risk of bradycardic events unless already treated with a permanent pacemaker

Ages: 50 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13885 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R Hiatt, MD, Study Chair — University of Colorado School of Medicine; Peter Held, MD, Study Director — AstraZeneca
Locations (585):
- United States (242):
  - Research Site, Alexander City, Alabama
  - Research Site, Auburn, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Cottonwood, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Berkeley, California
  - Research Site, Beverly Hills, California
  - Research Site, Chula Vista, California
  - Research Site, El Cajon, California
  - Research Site, Fresno, California
  - Research Site, La Jolla, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Mission Viejo, California
  - Research Site, Moreno Valley, California
  - Research Site, Northridge, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Palo Alto, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Loveland, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Guilford, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlantis, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hudson, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Plantation, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Stuart, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Trinity, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Wellington, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Lithonia, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Martinez, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Arlington Heights, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Rock Island, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Elkhart, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Edgewood, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Bossier City, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Beltsville, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Greenbelt, Maryland
  - Research Site, Fall River, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Flint, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Mount Clemens, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Belleville, New Jersey
  - Research Site, Bridgewater, New Jersey
  - Research Site, Camden, New Jersey
  - Research Site, East Orange, New Jersey
  - Research Site, Eatontown, New Jersey
  - Research Site, Elmer, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Freehold, New Jersey
  - Research Site, Hackensack, New Jersey
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Linden, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Ocean City, New Jersey
  - Research Site, Sewell, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, West Orange, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Hawthorne, New York
  - Research Site, Johnson City, New York
  - Research Site, Liverpool, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Saratoga Springs, New York
  - Research Site, The Bronx, New York
  - Research Site, Troy, New York
  - Research Site, Williamsville, New York
  - Research Site, Yonkers, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Minot, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hillsboro, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Dunmore, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Newport, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Wormleysburg, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greenwood, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Friendswood, Texas
  - Research Site, Houston, Texas
  - Research Site, Hurst, Texas
  - Research Site, Killeen, Texas
  - Research Site, Lubbock, Texas
  - Research Site, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Odessa, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Tyler, Texas
  - Research Site, Victoria, Texas
  - Research Site, Webster, Texas
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Leesburg, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Puyallup, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, South Charleston, West Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Manitowoc, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Wausau, Wisconsin
- Argentina (10):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudadela
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, Rosario Santa Fe
  - Research Site, San Nicolás
  - Research Site, Santa Fe
- Brazil (15):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Campinas
  - Research Site, Canoas
  - Research Site, Curitiba
  - Research Site, Juiz de Fora
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Bernardo do Campo
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Tatuí
  - Research Site, Uberlândia
- Bulgaria (12):
  - Research Site, Burgas
  - Research Site, Gotse Delchev
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Razlog
  - Research Site, Rousse
  - Research Site, Samokov
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Sofia
- Canada (19):
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Bridgewater, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Brossard, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Chicoutimi
- Chile (5):
  - Research Site, Concepción
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (13):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Fuzhou
  - Research Site, Haerbin
  - Research Site, Hubei
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
- Czechia (11):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Jindřichův Hradec
  - Research Site, Kladno
  - Research Site, Liberec
  - Research Site, Olomouc
  - Research Site, Ostrava-Dubina
  - Research Site, Prague
  - Research Site, Slaný
- France (22):
  - Research Site, Amiens
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Castelnau-le-Lez
  - Research Site, Dijon
  - Research Site, La Tronche
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Limoges
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Rambouillet
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Thionville
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Ettlingen
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kaiserslautern
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Merseburg
  - Research Site, München
  - Research Site, Riesa
  - Research Site, Tübingen
  - Research Site, Wesel
- Hungary (16):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gyöngyös
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Szombathely
  - Research Site, Veszprém
- Italy (20):
  - Research Site, Ancona
  - Research Site, Avellino
  - Research Site, Castelfranco Veneto
  - Research Site, Catania
  - Research Site, Chieti
  - Research Site, Genova
  - Research Site, Lecce
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Oristano
  - Research Site, Padua
  - Research Site, Palermo
  - Research Site, Perugia
  - Research Site, Piacenza
  - Research Site, Pisa
  - Research Site, Ragusa
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo
  - Research Site, Siena
- Japan (32):
  - Research Site, Asahi-shi
  - Research Site, Beppu-shi
  - Research Site, Fukuoka
  - Research Site, Hamada-shi
  - Research Site, Himeji-shi
  - Research Site, Imabari
  - Research Site, Itabashi-ku
  - Research Site, Kasuga-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Koriyama-shi
  - Research Site, Kyoto
  - Research Site, Matsubara-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Mito
  - Research Site, Miura-gun
  - Research Site, Ogori-shi
  - Research Site, Ōita
  - Research Site, Sakaide-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Suwa-shi
  - Research Site, Toyonaka-shi
  - Research Site, Tsu
  - Research Site, Uji-shi
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yatsushiro-shi
  - Research Site, Yokohama
  - Research Site, Yokosuka-shi
- Mexico (10):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monclova
  - Research Site, Monterrey
  - Research Site, Querétaro
  - Research Site, San Luis Potosí City
  - Research Site, Tijuana
- Netherlands (9):
  - Research Site, Amsterdam
  - Research Site, Capelle aan den IJssel
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Heerlen
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Utrecht
- Philippines (13):
  - Research Site, Cebu
  - Research Site, Cebu City
  - Research Site, City of Taguig
  - Research Site, Dasmariñas
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Makati
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
  - Research Site, Tanauan
  - Research Site, Vigan
- Poland (15):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrów Mazowiecka
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zamość
  - Research Site, Łęczna
- Romania (13):
  - Research Site, Bacau
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Suceava
  - Research Site, Tg. Mures
  - Research Site, Timișoara
- Russia (15):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Gatchina
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Vladikavkaz
  - Research Site, Yekaterinburg
- Slovakia (8):
  - Research Site, Dunajská Streda
  - Research Site, Košice
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Trnava
  - Research Site, Žilina
- South Korea (8):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheonan-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (22):
  - Research Site, A Coruña
  - Research Site, Albacete
  - Research Site, Alcorcón
  - Research Site, Alicante
  - Research Site, Badalona (Barcelona)
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Boadilla del Monte
  - Research Site, Getafe
  - Research Site, Granada
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Huelva
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Mallorca
  - Research Site, Manises
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Sabadell
  - Research Site, Tarragona
  - Research Site, Toledo
  - Research Site, Valencia
- Sweden (9):
  - Research Site, Eksjö
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Karlstad
  - Research Site, Malmo
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Västerås
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Muang
  - Research Site, Songkhla
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Malatya
- Ukraine (7):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- United Kingdom (12):
  - Research Site, Aberdeen
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Cambridge
  - Research Site, Cheltenham
  - Research Site, Dundee
  - Research Site, Hull
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Worcester
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

REFERENCES:
- [Derived] Szarek M, Hess C, Patel MR, Jones WS, Berger JS, Baumgartner I, Katona B, Mahaffey KW, Norgren L, Blomster J, Rockhold FW, Hsia J, Fowkes FGR, Bonaca MP. Total Cardiovascular and Limb Events and the Impact of Polyvascular Disease in Chronic Symptomatic Peripheral Artery Disease. J Am Heart Assoc. 2022 Jun 7;11(11):e025504. doi: 10.1161/JAHA.122.025504. Epub 2022 May 27. PMID 35621222
- [Derived] Govsyeyev N, Nehler MR, Low Wang CC, Kavanagh S, Hiatt WR, Long C, Jones WS, Fowkes FGR, Berger JS, Baumgartner I, Patel MR, Goodney PP, Beckman JA, Katona BG, Mahaffey KW, Blomster J, Norgren L, Bonaca MP. Etiology and outcomes of amputation in patients with peripheral artery disease in the EUCLID trial. J Vasc Surg. 2022 Feb;75(2):660-670.e3. doi: 10.1016/j.jvs.2021.08.096. Epub 2021 Sep 28. PMID 34597783
- [Derived] Norgren L, North R, Baumgartner I, Berger JS, Blomster JI, Hiatt WR, Jones WS, Katona BG, Mahaffey KW, Mulder H, Patel MR, Rockhold FW, Fowkes FGR. World regional differences in outcomes for patients with peripheral artery disease: Insights from the EUCLID trial. Vasc Med. 2022 Feb;27(1):21-29. doi: 10.1177/1358863X211038620. Epub 2021 Sep 13. PMID 34516308
- [Derived] Hiatt WR, Hess CN, Bonaca MP, Kavanagh S, Patel MR, Baumgartner I, Berger JS, Blomster JI, Jones WS, Katona BG, Mahaffey KW, Norgren L, Rockhold FW, Fowkes FGR. Ankle-Brachial Index for Risk Stratification in Patients With Symptomatic Peripheral Artery Disease With and Without Prior Lower Extremity Revascularization: Observations From the EUCLID Trial. Circ Cardiovasc Interv. 2021 Jul;14(7):e009871. doi: 10.1161/CIRCINTERVENTIONS.120.009871. Epub 2021 Jul 13. PMID 34253048
- [Derived] Hsia J, Kavanagh ST, Hopley CW, Baumgartner I, Berger JS, Fowkes GR, Jones WS, Mahaffey KW, Norgren L, Patel MR, Rockhold F, Blomster J, Katona BG, Hiatt WR, Bonaca MP. Impact of chronic kidney disease on hemoglobin among patients with peripheral artery disease treated with P2Y12 inhibitors: Insights from the EUCLID trial. Vasc Med. 2021 Dec;26(6):608-612. doi: 10.1177/1358863X211017641. Epub 2021 Jun 3. PMID 34082620
- [Derived] Galani J, Mulder H, Rockhold FW, Weissler EH, Baumgartner I, Berger JS, Blomster JI, Fowkes FGR, Hiatt WR, Katona BG, Norgren L, Mahaffey KW, Quint JK, Patel MR, Jones WS. Association of Chronic Obstructive Pulmonary Disease with Morbidity and Mortality in Patients with Peripheral Artery Disease: Insights from the EUCLID Trial. Int J Chron Obstruct Pulmon Dis. 2021 Mar 29;16:841-851. doi: 10.2147/COPD.S292978. eCollection 2021. PMID 33824584
- [Derived] Kochar A, Mulder H, Rockhold FW, Baumgartner I, Berger JS, Blomster JI, Fowkes FGR, Katona BG, Lopes RD, Al-Khalidi HR, Mahaffey KW, Norgren L, Hiatt WR, Patel MR, Jones WS. Cause of Death Among Patients With Peripheral Artery Disease: Insights From the EUCLID Trial. Circ Cardiovasc Qual Outcomes. 2020 Nov;13(11):e006550. doi: 10.1161/CIRCOUTCOMES.120.006550. Epub 2020 Nov 12. PMID 33176462
- [Derived] Gutierrez JA, Heizer GM, Jones WS, Rockhold FW, Mahaffey KW, Fowkes FGR, Berger JS, Baumgartner I, Held P, Katona BG, Norgren L, Blomster JI, Hiatt WR, Patel MR. CYP2C19 status and risk of major adverse cardiovascular events in peripheral artery disease: Insights from the EUCLID Trial. Am Heart J. 2020 Nov;229:118-120. doi: 10.1016/j.ahj.2020.07.017. Epub 2020 Aug 16. No abstract available. PMID 32950849
- [Derived] Fudim M, Hopley CW, Huang Z, Kavanagh S, Rockhold FW, Baumgartner I, Berger JS, Blomster JI, Fowkes FGR, Katona BG, Mahaffey KW, Norgren L, Ostrom C, Patel MR, Jones WS, Hiatt WR. Association of Hypertension and Arterial Blood Pressure on Limb and Cardiovascular Outcomes in Symptomatic Peripheral Artery Disease: The EUCLID Trial. Circ Cardiovasc Qual Outcomes. 2020 Sep;13(9):e006512. doi: 10.1161/CIRCOUTCOMES.120.006512. Epub 2020 Aug 31. PMID 32862697
- [Derived] Long CA, Mulder H, Fowkes FGR, Baumgartner I, Berger JS, Katona BG, Mahaffey KW, Norgren L, Blomster JI, Rockhold FW, Hiatt WR, Patel MR, Jones WS, Nehler MR. Incidence and Factors Associated With Major Amputation in Patients With Peripheral Artery Disease: Insights From the EUCLID Trial. Circ Cardiovasc Qual Outcomes. 2020 Jul;13(7):e006399. doi: 10.1161/CIRCOUTCOMES.119.006399. Epub 2020 Jul 3. PMID 32615798
- [Derived] Haine A, Kavanagh S, Berger JS, Hess CN, Norgren L, Fowkes FGR, Katona BG, Mahaffey KW, Blomster JI, Patel MR, Jones WS, Rockhold FW, Hiatt WR, Baumgartner I; International Steering Committee and Investigators of the EUCLID Trial. Sex-Specific Risks of Major Cardiovascular and Limb Events in Patients With Symptomatic Peripheral Artery Disease. J Am Coll Cardiol. 2020 Feb 18;75(6):608-617. doi: 10.1016/j.jacc.2019.11.057. PMID 32057375
- [Derived] Ward R, Huang Z, Rockhold FW, Baumgartner I, Berger JS, Blomster JI, Fowkes FGR, Katona BG, Mahaffey KW, Norgren L, Vemulapalli S, Povsic TJ, Mehta R, Hiatt WR, Patel MR, Jones WS. Major bleeding in patients with peripheral artery disease: Insights from the EUCLID trial. Am Heart J. 2020 Feb;220:51-58. doi: 10.1016/j.ahj.2019.11.007. Epub 2019 Nov 18. PMID 31783279
- [Derived] Hopley CW, Kavanagh S, Patel MR, Ostrom C, Baumgartner I, Berger JS, Blomster JI, Fowkes FGR, Jones WS, Katona BG, Mahaffey KW, Norgren L, Rockhold FW, Hiatt WR. Chronic kidney disease and risk for cardiovascular and limb outcomes in patients with symptomatic peripheral artery disease: The EUCLID trial. Vasc Med. 2019 Oct;24(5):422-430. doi: 10.1177/1358863X19864172. Epub 2019 Jul 24. PMID 31339474
- [Derived] Hess CN, Huang Z, Patel MR, Baumgartner I, Berger JS, Blomster JI, Fowkes FGR, Held P, Jones WS, Katona B, Mahaffey KW, Norgren L, Rockhold FW, Hiatt WR. Acute Limb Ischemia in Peripheral Artery Disease. Circulation. 2019 Aug 13;140(7):556-565. doi: 10.1161/CIRCULATIONAHA.119.039773. Epub 2019 Jun 26. PMID 31238713
- [Derived] Kolls BJ, Sapp S, Rockhold FW, Jordan JD, Dombrowski KE, Fowkes FGR, Mahaffey KW, Berger JS, Katona BG, Blomster JI, Norgren L, Abramson BL, Leiva-Pons JL, Prieto JC, Sokurenko G, Hiatt WR, Jones WS, Patel MR. Stroke in Patients With Peripheral Artery Disease. Stroke. 2019 Jun;50(6):1356-1363. doi: 10.1161/STROKEAHA.118.023534. Epub 2019 May 16. PMID 31092165
- [Derived] Low Wang CC, Blomster JI, Heizer G, Berger JS, Baumgartner I, Fowkes FGR, Held P, Katona BG, Norgren L, Jones WS, Lopes RD, Olin JW, Rockhold FW, Mahaffey KW, Patel MR, Hiatt WR; EUCLID Trial Executive Committee and Investigators. Cardiovascular and Limb Outcomes in Patients With Diabetes and Peripheral Artery Disease: The EUCLID Trial. J Am Coll Cardiol. 2018 Dec 25;72(25):3274-3284. doi: 10.1016/j.jacc.2018.09.078. PMID 30573030
- [Derived] Olivier CB, Mulder H, Hiatt WR, Jones WS, Fowkes FGR, Rockhold FW, Berger JS, Baumgartner I, Held P, Katona BG, Norgren L, Blomster J, Patel MR, Mahaffey KW. Incidence, Characteristics, and Outcomes of Myocardial Infarction in Patients With Peripheral Artery Disease: Insights From the EUCLID Trial. JAMA Cardiol. 2019 Jan 1;4(1):7-15. doi: 10.1001/jamacardio.2018.4171. PMID 30540355
- [Derived] Baumgartner I, Norgren L, Fowkes FGR, Mulder H, Patel MR, Berger JS, Jones WS, Rockhold FW, Katona BG, Mahaffey K, Hiatt WR; Executive Committee and Investigators of the EUCLID Trial. Cardiovascular Outcomes After Lower Extremity Endovascular or Surgical Revascularization: The EUCLID Trial. J Am Coll Cardiol. 2018 Oct 2;72(14):1563-1572. doi: 10.1016/j.jacc.2018.07.046. PMID 30261955
- [Derived] Berger JS, Abramson BL, Lopes RD, Heizer G, Rockhold FW, Baumgartner I, Fowkes FGR, Held P, Katona BG, Norgren L, Jones WS, Millegard M, Blomster J, Reist C, Hiatt WR, Patel MR, Mahaffey KW. Ticagrelor versus clopidogrel in patients with symptomatic peripheral artery disease and prior coronary artery disease: Insights from the EUCLID trial. Vasc Med. 2018 Dec;23(6):523-530. doi: 10.1177/1358863X18775594. Epub 2018 Jul 11. PMID 29992857
- [Derived] Norgren L, Patel MR, Hiatt WR, Wojdyla DM, Fowkes FGR, Baumgartner I, Mahaffey KW, Berger JS, Jones WS, Katona BG, Held P, Blomster JI, Rockhold FW, Bjorck M; EUCLID Steering Committee and Investigators. Outcomes of Patients with Critical Limb Ischaemia in the EUCLID Trial. Eur J Vasc Endovasc Surg. 2018 Jan;55(1):109-117. doi: 10.1016/j.ejvs.2017.11.006. Epub 2017 Dec 20. PMID 29273390
- [Derived] Hiatt WR, Fowkes FG, Heizer G, Berger JS, Baumgartner I, Held P, Katona BG, Mahaffey KW, Norgren L, Jones WS, Blomster J, Millegard M, Reist C, Patel MR; EUCLID Trial Steering Committee and Investigators. Ticagrelor versus Clopidogrel in Symptomatic Peripheral Artery Disease. N Engl J Med. 2017 Jan 5;376(1):32-40. doi: 10.1056/NEJMoa1611688. Epub 2016 Nov 13. PMID 27959717
- [Derived] Jones WS, Baumgartner I, Hiatt WR, Heizer G, Conte MS, White CJ, Berger JS, Held P, Katona BG, Mahaffey KW, Norgren L, Blomster J, Millegard M, Reist C, Patel MR, Fowkes FG; International Steering Committee and Investigators of the EUCLID Trial. Ticagrelor Compared With Clopidogrel in Patients With Prior Lower Extremity Revascularization for Peripheral Artery Disease. Circulation. 2017 Jan 17;135(3):241-250. doi: 10.1161/CIRCULATIONAHA.116.025880. Epub 2016 Nov 13. PMID 27840336
- [Derived] Held P, Himmelmann A, Ditmarsch M. Ticagrelor for the treatment of atherosclerotic disease: insights from the PARTHENON clinical development program. Future Cardiol. 2016 Jul;12(4):405-18. doi: 10.2217/fca-2016-0028. Epub 2016 May 10. PMID 27160944
- See also: Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=491&filename=Redacted_Protocol.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 821 centres randomising patients across 28 countries. The first patient was enrolled on 04 December 2012. The last visit of the last patient took place on 26 September 2016. In total, 16237 patients were screened.
Pre-assignment Details: Screened patients randomised to study drug: 85.5%; n=13885 Patients who were not randomised: 14.5%; n=2352 Patients with inclusion criteria for symptomatic lower extremity PAD failed: n=489 Patients with poor metabolizer status for CYP2C19: n=616 Patients with other reason: n=1374
Period: Overall Study
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Started | 6930 | 6955
Completed | 6807 (Includes patients who did not withdraw informed consent prior to the PACD) | 6842 (Includes patients who did not withdraw informed consent prior to the PACD)
Not Completed | 123 | 113
Not completed — Withdrawal by Subject | 123 | 113

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 90mg bd | Clopidogrel 75mg od | Total
Number analyzed (Participants) | 6930 | 6955 | 13885
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 66.6 (8.4) | 66.5 (8.5) | 66.6 (8.4)
Age, Customized [Number; unit: Participants]
  <65 years | 2900 | 2985 | 5885
  Between 65 and 75 years | 2925 | 2850 | 5775
  >75 years | 1105 | 1120 | 2225
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1908 | 1980 | 3888
  Male | 5022 | 4975 | 9997
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic Or Latino | 1046 | 1067 | 2113
  Not Hispanic Or Latino | 5884 | 5888 | 11772
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian Or Alaska Native | 63 | 62 | 125
  Asian | 824 | 810 | 1634
  Black Or African American | 280 | 289 | 569
  Native Hawaiian Or Other Pacific Islander | 2 | 3 | 5
  Other | 110 | 132 | 242
  White | 5651 | 5659 | 11310

OUTCOME MEASURES:

1. Primary Outcome: Composite of Cardiovascular (CV) Death/MI/Ischemic Stroke
Description: Participants with CV death, myocardial infarction (MI) or ischemic stroke. If no event, censoring occurs at the minimum of (primary analysis censoring date (PACD), last endpoint assessment date, non-CV death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participants | 751 | 740
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.650, Regression, Cox — The hypothesis will be tested at the 4.94% two-sided significance level to account for the planned interim analysis with the overall type I error preserved at 5%. A hierarchical test sequence will be used to address the issue of multiple testing; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.92 to 1.13]

2. Secondary Outcome: Composite of CV Death, MI, Ischemic Stroke, and ALI
Description: Participants with CV death, MI, ischemic stroke or acute limb ischemia (ALI). If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, non-CV death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 839 | 833
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.738, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.92 to 1.12]

3. Secondary Outcome: CV Death
Description: Participants with CV death. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, non-CV death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 363 | 343
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.400, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.92 to 1.23]

4. Secondary Outcome: MI
Description: Participants with MI. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 349 | 334
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.482, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.91 to 1.23]

5. Secondary Outcome: All-cause Mortality
Description: Participants with all-cause death. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 628 | 635
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.913, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.89 to 1.11]

6. Secondary Outcome: Composite of CV Death, MI, and All-cause Stroke (Ischemic or Hemorrhagic)
Description: Participants with CV death, MI or all-cause stroke. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, non-CV death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 766 | 759
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.724, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.92 to 1.13]

7. Secondary Outcome: ALI
Description: Participants with ALI. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 117 | 115
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.846, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.79 to 1.33]

8. Secondary Outcome: Lower Extremity Revascularization
Description: Participants with lower extremity revascularization (LER). If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 846 | 892
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.298, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.87 to 1.05]

9. Secondary Outcome: Any Revascularisation (Coronary, Peripheral [Limb, Mesenteric, Renal, Carotid and Other])
Description: Participants with any revascularization. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 1211 | 1250
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.462, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.90 to 1.05]

10. Other Pre Specified Outcome: Net Clinical Benefit (Composite of CV Death/MI/Ischemic Stroke/Fatal Bleeding/Intracranial Bleeding)
Description: Participants with CV death, MI, ischemic stroke, fatal bleeding or intracranial bleeding. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, non-CV death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 789 | 786
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.793, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.92 to 1.12]

11. Other Pre Specified Outcome: Net Clinical Benefit (Composite of All-cause Mortality/MI/Ischemic Stroke/Fatal Bleeding/Intracranial Bleeding)
Description: Participants with all-cause death, MI, ischemic stroke, fatal bleeding or intracranial bleeding. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 983 | 992
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 1.000, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.92 to 1.09]

12. Other Pre Specified Outcome: Net Clinical Benefit (Composite of All-cause Mortality/MI/Ischemic Stroke/ALI/Major Amputation/Fatal Bleeding/Intracranial Bleeding)
Description: Participants with all-cause death, MI, ischemic stroke, ALI, major amputation, fatal bleeding or intracranial bleeding. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 1119 | 1140
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.829, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.91 to 1.08]

13. Other Pre Specified Outcome: Net Clinical Benefit (Composite of All-cause Mortality/MI/Ischemic Stroke/ALI/Major Amputation/TIMI Major Bleeding)
Description: Participants with all-cause death, MI, ischemic stroke, ALI, major amputation or Thrombolysis in Myocardial Infarction (TIMI) major bleeding. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 1183 | 1199
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.949, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.92 to 1.08]

14. Other Pre Specified Outcome: Non-CV Death
Description: Participants with non-CV death. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, CV death)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 250 | 272
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.377, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.78 to 1.10]

15. Other Pre Specified Outcome: Changes in Fontaine Stage
Description: Progression of the clinical/symptomatic status of the limb by changes in Fontaine stage.
  Stage I - Asymptomatic Stage IIa - Intermittent claudication after more than 200 meters of pain free walking Stage IIb - Intermittent claudication after less than 200 meters of walking Stage III - Rest pain Stage IV - Ischemic ulcers or gangrene
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Groups:
- Ticagrelor - Stage I; Clopidogrel - Stage I: Baseline Fontaine stage I
- Ticagrelor - Stage IIa; Clopidogrel - Stage IIa: Baseline Fontaine stage IIa
- Ticagrelor - Stage IIb; Clopidogrel - Stage IIb: Baseline Fontaine stage IIb
- Ticagrelor - Stage III; Clopidogrel - Stage III: Baseline Fontaine stage III
- Ticagrelor - Stage IV; Clopidogrel - Stage IV: Baseline Fontaine stage IV
Arm/Group | Ticagrelor - Stage I | Ticagrelor - Stage IIa | Ticagrelor - Stage IIb | Ticagrelor - Stage III | Ticagrelor - Stage IV | Clopidogrel - Stage I | Clopidogrel - Stage IIa | Clopidogrel - Stage IIb | Clopidogrel - Stage III | Clopidogrel - Stage IV
Number analyzed (Participants) | 1309 | 3674 | 1620 | 186 | 140 | 1292 | 3736 | 1608 | 192 | 125
Participant
  Stage I - End of treatment | 775 | 683 | 171 | 15 | 26 | 743 | 723 | 198 | 33 | 19
  Stage IIa - End of treatment | 227 | 1948 | 560 | 41 | 28 | 230 | 1956 | 557 | 33 | 21
  Stage IIb - End of treatment | 45 | 269 | 469 | 39 | 19 | 56 | 311 | 450 | 38 | 15
  Stage III - End of treatment | 7 | 24 | 12 | 31 | 7 | 9 | 15 | 23 | 23 | 12
  Stage IV - End of treatment | 7 | 7 | 5 | 1 | 13 | 4 | 7 | 10 | 5 | 13
  Missing - End of treatment | 248 | 743 | 403 | 59 | 47 | 250 | 724 | 370 | 60 | 45

16. Other Pre Specified Outcome: Changes in Rutherford Classification
Description: Progression of the clinical/symptomatic status of the limb by changes in Rutherford classification.
  Category 0 - Asymptomatic Category 1 - Mild claudication Category 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Category 3 - Severe claudication Category 4 - Rest pain Category 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Category 6 - Severe ischemic ulcers or frank gangrene
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Groups:
- Ticagrelor - Cat 0; Clopidogrel - Cat 0: Baseline Rutherford category 0
- Ticagrelor - Stage II; Clopidogrel - Cat 1/2: Baseline Rutherford category 1/2
- Ticagrelor - Cat 3; Clopidogrel - Cat 3: Baseline Rutherford category 3
- Ticagrelor - Cat 4; Clopidogrel - Cat 4: Baseline Rutherford category 4
- Ticagrelor - Cat 5; Clopidogrel - Cat 5: Baseline Rutherford category 5
- Ticagrelor - Cat 6; Clopidogrel - Cat 6: Baseline Rutherford category 6
Arm/Group | Ticagrelor - Cat 0 | Ticagrelor - Stage II | Ticagrelor - Cat 3 | Ticagrelor - Cat 4 | Ticagrelor - Cat 5 | Ticagrelor - Cat 6 | Clopidogrel - Cat 0 | Clopidogrel - Cat 1/2 | Clopidogrel - Cat 3 | Clopidogrel - Cat 4 | Clopidogrel - Cat 5 | Clopidogrel - Cat 6
Number analyzed (Participants) | 1309 | 3674 | 1620 | 186 | 107 | 33 | 1292 | 3736 | 1608 | 192 | 100 | 25
Participant
  Category 0 - End of treatment | 775 | 683 | 171 | 15 | 23 | 3 | 743 | 723 | 198 | 33 | 13 | 6
  Category 1/2 - End of treatment | 227 | 1948 | 560 | 41 | 23 | 5 | 230 | 1956 | 557 | 33 | 18 | 3
  Category 3 - End of treatment | 45 | 269 | 469 | 39 | 13 | 6 | 56 | 311 | 450 | 38 | 12 | 3
  Category 4 - End of treatment | 7 | 24 | 12 | 31 | 4 | 3 | 9 | 15 | 23 | 23 | 11 | 1
  Category 5 - End of treatment | 5 | 4 | 3 | 1 | 11 | 0 | 2 | 6 | 6 | 4 | 12 | 1
  Category 6 - End of treatment | 2 | 3 | 2 | 0 | 0 | 2 | 2 | 1 | 4 | 1 | 0 | 0
  Missing - End of treatment | 248 | 743 | 403 | 59 | 33 | 14 | 250 | 724 | 370 | 60 | 34 | 11

17. Other Pre Specified Outcome: Change in ABI/TBI From Baseline
Description: Change in ankle brachial index (ABI) / toe brachial index (TBI).
  Ankle brachial index (ABI) is the ratio of blood pressures from the ankle and arm and is used for diagnosing peripheral arterial occlusive disease (PAOD):
  Normal: 1 to 1.29 Borderline: 0.91 to 0.99 Mild PAOD: 0.71 to 0.90 Medium severe PAOD: 0.41 to 0.7 Severe PAOD: <0.4
  Toe brachial index (TBI) is the ratio between the toe pressure and the higher brachial pressure, used for diagnosing PAOD when the ABI cannot be used:
  Normal: >0.7 Mild: 0.5-0.7 Moderate: 0.35-0.5 Moderate-Severe: <0.35 and toe pressure 40 mmHg Severe: <0.35 and toe pressure < 30 mmHg
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Mean (Standard Deviation); unit: Change in ABI/TBI
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6908 | 6940
Change in ABI/TBI
  ABI - 6 months N = 6184(Tica), 6319(Clopi) | 0.016 (0.136) | 0.011 (0.134)
  ABI - End of treatment N = 4951(Tica), 5073(Clopi) | 0.022 (0.167) | 0.016 (0.167)
  TBI - 6 months N = 55(Tica), 48(Clopi) | 0.050 (0.132) | 0.036 (0.137)
  TBI - End of treatment N = 36(Tica), 21(Clopi) | 0.059 (0.115) | -0.065 (0.304)

18. Other Pre Specified Outcome: Any Amputation Caused by PAD
Description: Participants with any amputation caused by peripheral arterial disease (PAD). If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 179 | 208
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.164, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.71 to 1.06]

19. Other Pre Specified Outcome: Major Amputation Caused by PAD
Description: Participants with major amputation caused by PAD. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 100 | 116
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.306, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.67 to 1.14]

20. Other Pre Specified Outcome: CV-related Hospitalization
Description: Participants with hospitalization associated with CV death, hospitalization due to MI, ischemic stroke, lower extremity revascularization, major amputation due to PAD, transient ischemic attack (TIA), coronary revascularization or unstable angina. If no event, censoring occurs at the minimum of (PACD, last endpoint assessment date, death date)
Time Frame: From randomization to PACD, an average of 2.5 years
Population: The population was the full analysis set, which included all randomized patients
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6930 | 6955
Participant | 1312 | 1314
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.887, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.93 to 1.09]

21. Other Pre Specified Outcome: TIMI Major Bleeding Events
Description: Participants with TIMI major bleeding event. If no event, censoring occurs at the minimum of (last endpoint assessment date, death date, 7 days after last dose of study drug)
Time Frame: From the date of first dose and up to and including 7 days following the date of last dose of study drug
Population: The population was the safety analysis set, which included all patients who received at least 1 dose of randomized ticagrelor or clopidogrel and for whom post-dose data are available
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6910 | 6932
Participant | 113 | 109
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.489, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.84 to 1.43]

22. Other Pre Specified Outcome: TIMI Major or Minor Bleeding Events
Description: Participants with TIMI major or minor bleeding event. If no event, censoring occurs at the minimum of (last endpoint assessment date, death date, 7 days after last dose of study drug)
Time Frame: From the date of first dose and up to and including 7 days following the date of last dose of study drug
Population: as for outcome 21
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6910 | 6932
Participant | 193 | 175
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.138, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.95 to 1.43]

23. Other Pre Specified Outcome: PLATO Major Bleeding Events
Description: Participants with PLATO major bleeding event. If no event, censoring occurs at the minimum of (last endpoint assessment date, death date, 7 days after last dose of study drug)
Time Frame: From the date of first dose and up to and including 7 days following the date of last dose of study drug
Population: as for outcome 21
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6910 | 6932
Participant | 206 | 188
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p = 0.139, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.95 to 1.41]

24. Other Pre Specified Outcome: Premature Permanent Discontinuation of Study Drug Due to Any Bleeding Event
Description: Participants with a permanent discontinuation of study drug due to any bleeding event. If no event, censoring occurs at the minimum of (last endpoint assessment date, death date, 7 days after last dose of study drug)
Time Frame: From the date of first dose and up to and including 7 days following the date of last dose of study drug
Population: The population was the saftey analysis set, which included all patients who received at least 1 dose of randomized ticagrelor or clopidogrel and for whom post-dose data are available
Measure: Number; unit: Participant
Arm/Group | Ticagrelor 90 mg bd | Clopidogrel 75 mg od
Number analyzed (Participants) | 6910 | 6932
Participant | 168 | 112
Statistical Analysis 1: Comparison: Ticagrelor 90 mg bd vs Clopidogrel 75 mg od; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.58, 95% CI 2-sided [1.24 to 2.00]

ADVERSE EVENTS:
Time Frame: On or after the date of first dose and up to and including 7 days following the date of last dose of study medication
Arm/Group | Clopidogrel 75mg od | Ticagrelor 90mg bd
Serious Adverse Events (participants affected / at risk) | 1788/6932 | 1716/6910
Other Adverse Events (participants affected / at risk) | 989/6932 | 1682/6910
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 75mg od (N=6932) | Ticagrelor 90mg bd (N=6910)
Anaemia (Blood and lymphatic system disorders) | 38 (40) | 39 (43)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Angina pectoris (Cardiac disorders) | 18 (20) | 32 (34)
Angina unstable (Cardiac disorders) | 6 (8) | 10 (11)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 8 (8) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 67 (69) | 69 (69)
Atrial flutter (Cardiac disorders) | 6 (6) | 11 (12)
Atrial tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 6 (6)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 5 (5)
Bradyarrhythmia (Cardiac disorders) | 4 (4) | 9 (9)
Bradycardia (Cardiac disorders) | 8 (8) | 4 (4)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 23 (29) | 28 (30)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 6 (6) | 6 (7)
Cardiac failure congestive (Cardiac disorders) | 88 (108) | 68 (81)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Coronary artery disease (Cardiac disorders) | 4 (4) | 8 (8)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Heart valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 3 (3)
Ischaemic cardiomyopathy (Cardiac disorders) | 4 (4) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 5 (5) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 5 (5) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 4 (5) | 4 (6)
Tachyarrhythmia (Cardiac disorders) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 3 (3) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 5 (5) | 10 (12)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 9 (9)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 4 (4)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 14 (17) | 14 (15)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Diabetic retinopathy (Eye disorders) | 3 (3) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 4 (4) | 2 (3)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 6 (6) | 1 (1)
Retinal haemorrhage (Eye disorders) | 2 (3) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinoschisis (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 8 (10)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 8 (8)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acid peptic disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 6 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 3 (3) | 5 (5)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 5 (5) | 6 (6)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 10 (10) | 8 (12)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 38 (41) | 34 (39)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 4 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 10 (11)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 2 (2)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 22 (23) | 20 (21)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 15 (16) | 14 (15)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 5 (5)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 8 (8) | 8 (8)
Pancreatitis acute (Gastrointestinal disorders) | 9 (12) | 4 (4)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (3) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 6 (7) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 2 (2) | 2 (2)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Tongue dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 9 (9)
Volvulus (Gastrointestinal disorders) | 1 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 3 (3) | 3 (4)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 7 (8) | 9 (9)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Complication of device removal (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Drowning (General disorders) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 3 (3) | 0 (0)
Medical device site erosion (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 6 (6)
Non-cardiac chest pain (General disorders) | 37 (38) | 37 (40)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 5 (5)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vascular stent restenosis (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangiolitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 3 (4) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 8 (9) | 14 (14)
Cholecystitis acute (Hepatobiliary disorders) | 10 (10) | 11 (11)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 13 (13) | 14 (16)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fatty liver alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 5 (5)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Allergy to chemicals (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2)
Overlap syndrome (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 2 (2) | 1 (1)
Abscess of salivary gland (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 2 (2) | 3 (3)
Appendicitis (Infections and infestations) | 9 (9) | 5 (5)
Appendicitis perforated (Infections and infestations) | 2 (2) | 2 (2)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Atypical mycobacterial pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 4 (4)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bone abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 19 (19) | 23 (24)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Carbuncle (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 26 (28) | 27 (28)
Cholangitis infective (Infections and infestations) | 1 (1) | 1 (1)
Cholecystitis infective (Infections and infestations) | 2 (2) | 2 (2)
Chronic hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 8 (8) | 4 (4)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 3 (3)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Corynebacterium bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 3 (3)
Device related infection (Infections and infestations) | 6 (6) | 5 (5)
Diabetic foot infection (Infections and infestations) | 2 (3) | 2 (2)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 7 (7) | 6 (6)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 3 (3) | 1 (1)
Echinococciasis (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 4 (4) | 5 (5)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder empyema (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 13 (13) | 12 (13)
Gastroenteritis salmonella (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Graft infection (Infections and infestations) | 3 (3) | 5 (5)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 2 (2)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 8 (8)
Intervertebral discitis (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 3 (5)
Liver abscess (Infections and infestations) | 0 (0) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 7 (7)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 2 (2) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 9 (10) | 7 (7)
Osteomyelitis chronic (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 6 (6) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 164 (175) | 137 (141)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 6 (6)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (3) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 10 (10) | 4 (4)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 4 (4)
Pyelonephritis (Infections and infestations) | 4 (5) | 5 (5)
Pyelonephritis acute (Infections and infestations) | 3 (3) | 4 (4)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 21 (22) | 21 (21)
Septic shock (Infections and infestations) | 13 (14) | 11 (11)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Splenic abscess (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Tetanus (Infections and infestations) | 0 (0) | 1 (1)
Tracheostomy infection (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 3 (3)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (3)
Urethral stricture post infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 40 (48) | 32 (34)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 13 (15)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 3 (4)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 8 (10)
Femoral neck fracture (Injury, poisoning and procedural complications) | 11 (11) | 12 (12)
Femur fracture (Injury, poisoning and procedural complications) | 13 (13) | 11 (11)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 13 (13) | 12 (12)
Humerus fracture (Injury, poisoning and procedural complications) | 10 (10) | 5 (5)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Lumbosacral plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Multiple fractures (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 7 (7) | 14 (14)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 11 (12) | 8 (8)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Radiation fibrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 7 (7) | 8 (8)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (6)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 7 (7) | 9 (9)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Vascular graft complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (4)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Computerised tomogram thorax abnormal (Investigations) | 1 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 4 (4) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Salmonella test positive (Investigations) | 0 (0) | 1 (1)
Stool analysis abnormal (Investigations) | 0 (0) | 1 (1)
Thyroid function test abnormal (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 10 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 10 (12) | 14 (15)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 18 (22) | 11 (11)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (5) | 6 (6)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Gout (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (10) | 15 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 12 (14) | 17 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 6 (7)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic syndrome (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 15 (15) | 12 (12)
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 41 (45) | 40 (41)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 6 (6)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 8 (8)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 8 (8)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 6 (6)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 9 (9)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Disseminated large cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endometrial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 8 (8)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head and neck cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 5 (5)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 11 (11)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 8 (8)
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (22) | 27 (27)
Lung squamous cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Malignant middle ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Nonkeratinising carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 15 (15)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectosigmoid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 12 (12)
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell cancer of the renal pelvis and ureter recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vaginal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 2 (2) | 2 (2)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 2 (2)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 2 (2) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 60 (64) | 56 (58)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 4 (4)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 2 (2)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 4 (5) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 3 (3)
Drug withdrawal convulsions (Nervous system disorders) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 4 (4) | 3 (3)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 6 (6) | 4 (4)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 6 (6) | 5 (5)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Hemianopia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 3 (3)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 2 (2)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Internal carotid artery kinking (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 2 (2)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 3 (3)
Lumbosacral plexopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Post stroke epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 5 (5) | 5 (5)
Radial nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 1 (1) | 1 (1)
Radicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 7 (7) | 3 (3)
Sleep paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (3)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 7 (7) | 4 (4)
Syncope (Nervous system disorders) | 18 (18) | 26 (27)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 4 (4)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 3 (3)
Wernicke's encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 2 (2) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 3 (3) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 2 (2) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 8 (8) | 5 (10)
Drug abuse (Psychiatric disorders) | 1 (1) | 1 (2)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2) | 2 (2)
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 3 (3) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 32 (32) | 48 (52)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 13 (14) | 20 (23)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 10 (11) | 8 (8)
Haemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 6 (6) | 2 (2)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 5 (5) | 5 (7)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 2 (3)
Perinephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal aneurysm (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal arteriosclerosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 4 (4) | 5 (6)
Renal atrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal failure (Renal and urinary disorders) | 19 (19) | 14 (14)
Renal impairment (Renal and urinary disorders) | 7 (7) | 6 (6)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 4 (4)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 5 (6)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 13 (13) | 10 (10)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Peyronie's disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 17 (18)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (9)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 71 (100) | 87 (113)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 11 (11)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 18 (18)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (12)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 8 (9) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Subacute cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 2 (2)
Aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 12 (12) | 9 (9)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 2 (2)
Aortic dissection (Vascular disorders) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 12 (12) | 7 (7)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Aorto-duodenal fistula (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Behcet's syndrome (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic artery stenosis (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 11 (11) | 12 (12)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (2)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 8 (8) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 30 (32) | 20 (20)
Hypertensive crisis (Vascular disorders) | 9 (9) | 10 (10)
Hypertensive emergency (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 5 (6)
Hypovolaemic shock (Vascular disorders) | 3 (3) | 2 (2)
Iliac artery perforation (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 2 (2)
May-Thurner syndrome (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 5 (5) | 7 (7)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Renovascular hypertension (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 3 (3) | 4 (4)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 2 (2)
Thromboangiitis obliterans (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 3 (3)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein ruptured (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous perforation (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 3 (3)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 75mg od (N=6932) | Ticagrelor 90mg bd (N=6910)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 264 (289) | 817 (968)
Haemorrhage (Vascular disorders) | 787 (1078) | 997 (1451)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No